CLINICAL TRIAL: NCT06847204
Title: EFFICACY OF COLCHICINE IN IMPROVING CLINICAL OUTCOMES IN PATIENTS WITH MILD TO MODERATE COVID-19 PNEUMONIA IN LAHORE: A RANDOMIZED CONTROL TRIAL
Acronym: Colchicine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zaeema Kanwal (Other Government)
Responsible Party: Sponsor-Investigator, Zaeema Kanwal, Zkanwal, Lahore General Hospital
Organization: Lahore General Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: farahkchem@yahoo.com
Record Dates: First submitted 2025-02-24; First posted 2025-02-26 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-02

CONDITIONS: COVID - 19
MeSH Terms: conditions — COVID-19 | interventions — Colchicine; Tablets

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine group (Active Comparator): Experimental group will be given tab colchicine 0.5 mg 1 daily in addition to usual treatment for Covid-19 pneumonia mild , moderate cases.
  Interventions: Drug: Colchicine 0.5 MG Oral Tablet
- Controlled group (No Intervention): This group will only be given usual treatment for covid 19 pneumonia ( anti coagulation, steroid, nebulisation)

INTERVENTIONS:
Drug: Colchicine 0.5 MG Oral Tablet — Colchicine is anti inflammatory drug which will be given to Covid pneumonia patients and their benefit will be observed in them
  Arms: Colchicine group

SUMMARY:
This study is for patients suffering from COVID-19 pneumonia (mild to moderate cases) ; especially in developing countries where expensive drugs are not available.

Colchicine is an economically favourable anti inflammatory drug readily Used for gout patients but is being given experimentally in Covid 19 patients .

Study has been designed in this way that drug has been given carefully to patients on which there will be no to minimum side effects . It is only to see beneficial effects if any present in Covid pneumonia patients which will be observed by clinical & lab improvement.

DETAILED DESCRIPTION:
Colchicine, an anti-inflammatory drug used conventionally to treat gout and pericarditis. This study shows effectiveness of colchicine in enhancing clinical outcomes in mildly to moderately severe COVID-19 pneumonia patients.

Improvement will be observed in terms of shorter hospital admissions and oxygen dependency .

ELIGIBILITY:
Inclusion Criteria:

* Patients with laboratory-confirmed COVID-19 infection through a PCR test using a nasopharyngeal swab specimen, or the presence of at least two of the following four inflammatory criteria: C-reactive protein (CRP) level > 4 mg/dL, D-dimer level > 1 mg/L, ferritin level > 1000 ng/mL, along with fever ≥ 38 °C and respiratory distress Patients having supplemental oxygen requirement. Patients who provide informed consent to participate in the study. Patients having normal levels of serum Ca2+ and K+; QT interval <450 ms at 12 derivations ECG (Colchicine has been associated with potential cardiac side effects, including disturbances in electrolyte levels and QT interval prolongation. Normal levels of these electrolytes help minimise the risk of cardiac arrhythmias or other adverse events.

Exclusion Criteria:

Known hypersensitivity or allergy to colchicine or any of its excipients. Patients with an estimated glomerular filtration rate (eGFR) below 45 mL/min/1.73 m^2 or advanced liver disease (Child-Pugh Class B or C). Patients taking medications known to have significant interactions with colchicine, such as strong CYP3A4 inhibitors (e.g., clarithromycin, ketoconazole), P-glycoprotein inhibitors (e.g., cyclosporine), or medications associated with myelosuppression (e.g., azathioprine, cyclophosphamide). Patients with pre-existing medical conditions that, in the opinion of the investigator, could pose a significant risk or interfere with the interpretation of the study results (e.g., severe heart failure, uncontrolled arrhythmias, uncontrolled diabetes, or active malignancies).

Pregnant or lactating individuals. Patients deemed by the investigator to be in imminent danger of death or unlikely to survive the duration of study due to some other disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Hospital stay and oxygen dependence | Over a period of 07 days per patient after start of experimental drug
  Patients will be monitored for prolonged hospital stay and decrease /increase of oxygen requirement.

SECONDARY OUTCOMES:
Reduce levels of inflammatory markers | 7 days per patient
  There is a surge in inflammatory marker of Covid patients Their pattern will be monitored since the start of experimental medication and after 7 th day of medication.

CONTACTS AND LOCATIONS:
Locations (1):
- General hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided